CLINICAL TRIAL: NCT06776198
Title: Precision Therapy Based on Immune Microenvironment by Transcriptome Sequencing of Osteosarcoma, a Prospective, Multi-cohort Exploratory Clinical Study
Acronym: PTMTO
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Other Study IDs: PKUPH-sarcoma 21
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Osteosarcoma; Transcriptome; Tumor Microenvironment; Precision Medicine
Keywords: osteosarcoma; transcriptome; tumor microenviroment; precision medicine
MeSH Terms: conditions — Osteosarcoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Wholeexome sequencing (WES) and RNA sequencing (RNA-seq)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Immune-Enriched, Fibrotic Group (IE/F)
  Interventions: Drug: Chemotherapy
- Immune-Enriched, Non-Fibrotic Group (IE)
  Interventions: Drug: Chemotherapy
- Fibrotic Group (F)
  Interventions: Drug: Chemotherapy
- Depleted Group (D)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Group IE/F: After progression, try LRRC15 ADC + PD-1 inhibitors; Group IE: After progression, try simple anti-PD-1 inhibitors; Group F: After progression, try LRRC15 ADC; Group D: After progression, try B7-H3 ADC or other irrinotecan analogue

SUMMARY:
Bagaev et al. have identified four tumor microenvironment (TME) subtypes that are conserved across diverse cancers and correlated with immunotherapy response in melanoma, bladder, and gastric cancers. They provided a visual tool revealing the TME subtypes integrated with targetable genomic alterations, which provided a planetary view of each tumor that can aid in oncology clinical decision making. We aim to use this tool to prospectively analyse the biopsy specimens of osteosarcomas to identify their TME subtypes so as to deliver appropriate treatment strategy if these osteosarcomas experience disease progression afterwards. We will compare the past sequencing date stored in PKUPH bank so as to compare the event-free survival(EFS) of these patients to check the Superiority of this method later.

ELIGIBILITY:
Inclusion Criteria:

* (i) patients who have been suspected for osteosarcoma with enough clinical or radiographic information;
* (ii) patients who have evaluable lesions to resect or follow;
* (iii) patients who are planned to be operate with enough flesh specimens for this study.

Exclusion Criteria:

* (i) clinical information was not complete;
* (ii) lost to follow-up.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initially treated osteosarcoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | 2 year
  From biopsy to progression/last follow-up

SECONDARY OUTCOMES:
Event-free Survival (EFS) for the second time | 2 year
  From first progression to the second progression/last follow-up

OTHER OUTCOMES:
Correlation with some DNA target expression | 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagaev A, Kotlov N, Nomie K, Svekolkin V, Gafurov A, Isaeva O, Osokin N, Kozlov I, Frenkel F, Gancharova O, Almog N, Tsiper M, Ataullakhanov R, Fowler N. Conserved pan-cancer microenvironment subtypes predict response to immunotherapy. Cancer Cell. 2021 Jun 14;39(6):845-865.e7. doi: 10.1016/j.ccell.2021.04.014. Epub 2021 May 20. PMID 34019806